CLINICAL TRIAL: NCT07117539
Title: Impact of Laryngeal Mask Combined With Visual Bronchial Blocker on Pharyngolaryngeal Injuries After Pulmonary Resection
Brief Title: Impact of Different Lung Isolation Devices on Pharyngolaryngeal Injuries After Pulmonary Resection
Acronym: PLIAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tingting Li (Other)
Collaborators: Charta Foundation (Other)
Responsible Party: Sponsor-Investigator, Tingting Li, Attending physician, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: JRH000032
Record Dates: First submitted 2025-07-16; First posted 2025-08-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Neoplasm
Keywords: pulmonary resection; one-lung ventilation; pharyngolaryngeal injuries; lung isolation devices
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- visual bronchial blocker group（VBB） (Experimental): Laryngeal Mask Airway(LMA) size selection based on patient weight (≥70kg: size 5, 50-70kg: size 4, <50kg: size 3)；Standard LMA insertion technique in supine position；Visual bronchial blocker inserted through LMA central channel；Blocker advancement under direct vision to identify carina
  Interventions: Device: visual bronchial blocker (VBB)
- double-lumen endotracheal tube group（DLT） (Active Comparator): Size selection based on patient gender and height: Male: >180cm (37F), 160-180cm (35F), <160cm (32-35F)；Female: >160cm (35F), <155cm (32F), 155-160cm (individualized)；Standard laryngoscopy and DLT insertion；Fiberoptic bronchoscopy confirmation of positioning；Tracheal cuff pressure 25 cmH2O, bronchial cuff pressure 30 cmH2O
  Interventions: Device: double-lumen endotracheal tube (DLT)

INTERVENTIONS:
Device: visual bronchial blocker (VBB) — lung isolation with visual bronchial blocker
  Arms: visual bronchial blocker group（VBB）
Device: double-lumen endotracheal tube (DLT) — lung isolation with double-lumen endotracheal tube
  Arms: double-lumen endotracheal tube group（DLT）

SUMMARY:
The goal of this clinical trial is to assess the impact of laryngeal mask combined with visual bronchial blocker on pharyngolaryngeal injury after pulmonary resection in patients with pulmonary nodules. The main question it aims to answer is:

the incidence of postoperative pharyngolaryngeal injury within 24h : sore throat and hoarseness ? Researchers will compare the visual bronchial blocker group (VBB) with the double-lumen endotracheal tube group (DLT) to see if the visual bronchial blocker group can minimize laryngopharyngeal injury after pulmonary resection.

DETAILED DESCRIPTION:
Background: Video-assisted thoracoscopic surgery (VATS) necessitates effective lung isolation techniques. While double-lumen endotracheal tubes (DLT) remain the gold standard, they are associated with significant airway trauma and postoperative laryngopharyngeal morbidity. Laryngeal mask airway (LMA) combined with bronchial blockers represents a promising alternative; however, conventional bronchial blockers pose limitations including challenging positioning and potential airway injury. Novel visual bronchial blocker technology offers enhanced positioning accuracy and reduced airway manipulation, potentially minimizing laryngopharyngeal injury while maintaining effective lung isolation.

Objective: To compare the efficacy and safety of LMA combined with a visual bronchial blocker versus DLT for lung isolation in VATS, with a primary focus on reducing postoperative laryngopharyngeal injury.

Methods: This prospective, randomized, controlled, single-blind, multicenter clinical trial will enroll 270 patients scheduled for elective VATS anatomical lung resection. Participants will be randomly allocated (1:1 ratio) to either the visual bronchial blocker group (VBB group, n=135) or the DLT group (n=135) across three major thoracic surgery centers. The primary outcome is the incidence of laryngopharyngeal injury (sore throat and/or hoarseness) at 24 hours postoperatively. Secondary outcomes include laryngopharyngeal injury at 1 hour and 48 hours postoperatively, intraoperative device dislodgement, hypoxemia (SpO₂ < 90%), quality of lung collapse, airway instrumentation time, hemodynamic fluctuations, emergence quality, device-related complications, and hospital length of stay. Statistical analysis will be performed using SPSS 24.0, employing appropriate parametric and non-parametric tests.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Scheduled for elective VATS pulmonary resection under general anesthesia
* American Society of Anesthesiologists (ASA) physical status I-III
* Body mass index (BMI) 18.5-30.0 kg/m²
* Written informed consent

Exclusion Criteria:

* Anticipated difficult airway (Mallampati class IV, previous difficult intubation, airway abnormalities)
* Gastroesophageal reflux disease or gastric retention
* Active pulmonary infection or bleeding
* Severe pulmonary dysfunction (FEV1 <50% predicted)
* Previous lung surgery or bilateral lung surgery
* Cognitive impairment affecting outcome assessment
* Chronic throat pain or voice abnormalities within 24 hours preoperatively
* Abnormal right upper lobe bronchial anatomy on preoperative CT for right-sided procedures
* Any condition deemed unsuitable for study participation by anesthesiologist or surgeon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2025-08-18 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of pharyngolaryngeal injuries within postoperative 24 hours | within postoperative 24 hours
  sore throat and hoarseness

SECONDARY OUTCOMES:
Incidence of pharyngolaryngeal injuries within postoperative an hour | within postoperative an hour
  sore throat and hoarseness
Incidence of pharyngolaryngeal injuries within postoperative 48 hours | within postoperative 48 hours
  sore throat and hoarseness
Intraoperative device displacement | during the operation
  lung re-expansion, airway pressure changes
Intraoperative hypoxemia | during the operation
  SpO2 < 91%
Lung collapse quality | at 5, 10, and 20 minute during single-lung ventilation
  The Lung Collapse Scale (LCS) is a standardized tool used in thoracic surgery to evaluate the degree of lung deflation during procedures requiring single-lung ventilation.(A score of 0: No lung collapse ; A score of 8: Satisfactory lung collapse.; A score of 10: Complete lung collapse )
Intubation time | during anesthesia procedure
  from mouth opening to successful device placement
Hemodynamic changes | during anesthesia procedure
  blood pressure variations before and after intubation
Recovery quality: post-extubation cough | periprocedural (during anesthesia recovery)
  Post-extubation Cough Severity Scale (4-point Grading System) : Grade 0 (No cough); Grade 1( Mild cough: 1-2 episodes, duration <5 seconds ); Grade 2 (Moderate cough: 3-4 episodes, duration 5-15 seconds); Grade 3 (Severe cough ≥5 episodes, duration >15 seconds, with breath-holding and facial flushing)
Device-related complications | during the operation
  intraoperative displacement, air leak, repositioning requirements
Length of hospital stay | perioperative/periprocedural
  Surgery-to-Discharge Interval(SDI): measures the time from surgery end (e.g., leaving the operating room) to discharge.Assesses recovery efficiency and effectiveness of Enhanced Recovery After Surgery (ERAS) protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Jingxiang Wu, Study Director — Shanghai Chest Hospital; Tingting Li, Principal Investigator — Shanghai Chest Hospital
Locations (3):
- China (3):
  - Shanghai Chest Hospital, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - The Second Military Medical University Changhai Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Y, Li T, Wei J, Bao R, Lv X, Wang JF, Wu J. Laryngeal mask airway combined with visual bronchial blocker versus double-lumen tube for lung isolation in video-assisted thoracoscopic surgery: a protocol for a multicentre randomised controlled trial. BMJ Open. 2025 Dec 30;15(12):e110539. doi: 10.1136/bmjopen-2025-110539. PMID 41469076